CLINICAL TRIAL: NCT01144364
Title: A Randomized, Open-label Study of MabThera Maintenance Therapy Compared With no Further Therapy After a Brief Induction With Chemotherapy Plus MabThera on Failure-free Survival in Treatment-naïve Elderly Patients With Advanced Follicular Lymphoma
Brief Title: A Study of MabThera (Rituximab) in Elderly Patients With Untreated Follicular Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML17638
Record Dates: First submitted 2010-06-11; First posted 2010-06-15 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-06

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab [Mabthera/Rituxan]

INTERVENTIONS:
Drug: rituximab [Mabthera/Rituxan] — Intravenous repeating dose

SUMMARY:
This study will evaluate the efficacy and safety of brief induction therapy with a chemotherapeutic regimen containing MabThera, followed by either maintenance therapy with MabThera or no further therapy. The anticipated time on study treatment is 1-2 years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 60-75 years of age;
* B-cell follicular NHL;
* no previous treatment;
* active disease, with rapid progression.

Exclusion Criteria:

* other cancer within 3 years of study, except carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, or ductal carcinoma in situ of the breast treated with lumpectomy;
* long-term use (>1 month) of systemic corticosteroids;
* central nervous system involvement;
* history of significant cardiovascular disease;
* positive test result for HIV, or hepatitis B or C.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2004-01-19 (Actual); Primary Completion 2011-07-21 (Actual); Study Completion 2011-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (45):
- Italy (45):
  - Ospedale Civile Dello Spirito Santo; Divisione Di Ematologia, Pescara, Abruzzo
  - Uni Degli Studi Di Bari, Policlinico; Cattedra Di Ematologia,Dipart. Di Medicina Interna E Publica, Bari, Apulia
  - IRCCS Ospedale Casa Sollievo Della Sofferenza; Ematologia E Trapianto Di Midollo Osseo, San Giovanni Rotondo, Apulia
  - Ospedale Riuniti; Divisione Di Ematologia, Reggio Calabria, Calabria
  - Istituto Nazionale Tumori Irccs Fondazione g. Pascale;s.c. Ematologia Oncologica, Napoli, Campania
  - Nuovo Policlinico, Ii Facolta; Divisione Di Ematologia, Napoli, Campania
  - Ospedale Cardarelli; Divisione Di Ematologia, Napoli, Campania
  - Presidio Ospedaliero Umberto I; U.O. Di Medicina Interna Ed Oncoematologia, Nocera Inferiore, Campania
  - A.O. Universitaria Policlinico S.Orsola-Malpighi Di Bologna, Bologna, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Ematologia, Modena, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Radiologia, Modena, Emilia-Romagna
  - Az. Osp. Ospedale Civile; U.O. Di Oncologia Medica Ed Ematologia, Piacenza, Emilia-Romagna
  - Az. Osp. S. Maria Delle Croci; U.O. Di Ematologia, Ravenna, Emilia-Romagna
  - Az. Osp. Arcispedale S. Maria Nuova; U.O. Di Ematologia, Reggio Emilia, Emilia-Romagna
  - Policlinico Universitario; Clinica Oncologia - Padiglione Pennato, Udine, Friuli Venezia Giulia
  - Ospedale S. Eugenio; Divisione Di Ematologia, Rome, Lazio
  - Universita' Degli Studi La Sapienza-Ist.Di Ematologia;Dip. Biotecnologie Cel CELLULARI ED EMATOLOGIA, Rome, Lazio
  - Uni Cattolica; Divisione Di Ematologia, Rome, Lazio
  - ASST PAPA GIOVANNI XXIII; Ematologia, Bergamo, Lombardy
  - A.O. Spedali Civili Di Brescia-P.O. Spedali Civili;U.O. Ematologia, Brescia, Lombardy
  - ASST DI CREMONA; U.O.S. di Ematologia, Cremona, Lombardy
  - Ospedale Maggiore Di Milano; U.O. Ematologia I - Padiglione Marcora, Milan, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 1, Milan, Lombardy
  - Ist. Nazionale Per Lo Studio E Cura Dei Tumori; Div. Ematologia Trapianto Midollo Osseo Allogenico, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - ASST DI MONZA; Ematologia, Monza, Lombardy
  - Ospedale Civile SS. Antonio E Biagio DI Alessandria; Ematologia, Alessandria, Piedmont
  - Az. Osp. Di Biella; Divisione Di Ematologia, Biella, Piedmont
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo; Dipartimento Oncologico, Candiolo, Piedmont
  - Az. Osp. S. Croce Ospedale Generale; Sezione Di Ematologia, Cuneo, Piedmont
  - Az. Osp. S. Luigi Gonzaga; Malattie Apparato Respiratorio 5 Ad Indirizzo Oncologico, Orbassano, Piedmont
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino; Ematologia 1, Turin, Piedmont
  - A.O.U. Citta' Della Salute E Della Scienza-P.O. Molinette;S.C. Ematologia, Turin, Piedmont
  - Ospedale Oncologico A Businco-Cagliari; Ematologia Sez., Cagliari, Sardinia
  - Az. Osp. Papardo; Struttura Complessa Di Ematologia, Messina, Sicily
  - Ospedale V. Cervello; U.O. Ematologia E Trapianti, Palermo, Sicily
  - Ospedale Ferrarotto; Divisione Di Ematologia, Via S. Sofia 78, Sicily
  - Ospedale Regionale Di Torrette; Clinica Di Ematologia, Ancona, The Marches
  - Ospedale Civile; S.C. Ematologia, Pesaro, The Marches
  - Azienda Sanitaria Di Bolzano; Ematologia E Centro Trapianto Mid.Osseo, Bolzano, Trentino-Alto Adige
  - Az. Osp. Di Careggi; Divisione Di Ematologia, Florence, Tuscany
  - Ospedale Santa Chiara; Unita Operativa Di Ematologia, Pisa, Tuscany
  - Dept. Medicina Clinica E Sperimentale; Sez. Medicina Interna E Scienze Oncologiche - Pol. Monteluce, Perugia, Umbria
  - Ospedale Civile Ss. Giovanni E Paolo; Ematologia, Venezia, Veneto
  - Uni Di Verona Policlinico G.B. Rossi; Divisione E Cattedra Di Ematologia, Verona, Veneto

REFERENCES:
- [Derived] Ladetto M, Lobetti-Bodoni C, Mantoan B, Ceccarelli M, Boccomini C, Genuardi E, Chiappella A, Baldini L, Rossi G, Pulsoni A, Di Raimondo F, Rigacci L, Pinto A, Galimberti S, Bari A, Rota-Scalabrini D, Ferrari A, Zaja F, Gallamini A, Specchia G, Musto P, Rossi FG, Gamba E, Evangelista A, Vitolo U; Fondazione Italiana Linfomi. Persistence of minimal residual disease in bone marrow predicts outcome in follicular lymphomas treated with a rituximab-intensive program. Blood. 2013 Nov 28;122(23):3759-66. doi: 10.1182/blood-2013-06-507319. Epub 2013 Oct 1. PMID 24085766
- [Derived] Vitolo U, Ladetto M, Boccomini C, Baldini L, De Angelis F, Tucci A, Botto B, Chiappella A, Chiarenza A, Pinto A, De Renzo A, Zaja F, Castellino C, Bari A, Alvarez De Celis I, Evangelista A, Parvis G, Gamba E, Lobetti-Bodoni C, Ciccone G, Rossi G. Rituximab maintenance compared with observation after brief first-line R-FND chemoimmunotherapy with rituximab consolidation in patients age older than 60 years with advanced follicular lymphoma: a phase III randomized study by the Fondazione Italiana Linfomi. J Clin Oncol. 2013 Sep 20;31(27):3351-9. doi: 10.1200/JCO.2012.44.8290. Epub 2013 Aug 19. PMID 23960180

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction Phase-Immunochemotherapy Rituximab-FND (R-FND): Cycles 1 to 4: Participants received rituximab: 375 milligrams per square meter (mg/m^2) intravenously (IV) on Day 1*, fludarabine (F): 25 mg/m^2 IV on Days 2-4*, mitoxantrone (N): 10 mg/m^2 IV on Day 2*, dexamethasone (D) 10 mg IV (total dose) on Days 2-4*. Cycles were repeated every 28 days for a total of 4 cycles. *In Cycle 1, rituximab was given on Day 8 in order to avoid tumour lysis syndrome. Consequently, in Cycle 1, fludarabine and dexamethasone were given on Days 1, 2, and 3. Mitoxantrone was given on Day 1.
- Rituximab Induction, Rituximab Maintenance: Induction Phase Cycle 1 (4-week cycle): Participants received mitoxantrone 10 mg/m^2 IV on Day 1, fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 1-3, and rituximab 375 mg/m^2 on Day 8. Induction Phase Cycles 2-4 (4-week cycle): Participants received rituximab 375 mg/m^2 IV on Day 1, mitoxantrone 10 mg/m^2 IV on Day 2, and fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 2-4. One month after completion of the above 4 cycles, participants were evaluated for tumor response (clinical and molecular evaluation). Responding participants (no progressive disease) received rituximab 375 mg/m^2 IV once weekly for a total of 4 weeks (4 total doses). Maintenance Phase: 3 months after induction treatment (Month 9), participants who showed at least a partial response after induction treatment received rituximab 375 mg/m^2 IV on Day 1. Doses were repeated every 2 months for a total of 4 doses.
- Rituximab Induction, Observation Maintenance: Induction Phase Cycle 1 (4-week cycle): Participants received mitoxantrone 10 mg/m^2 IV on Day 1, fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 1-3, and rituximab 375 mg/m^2 on Day 8. Induction Phase Cycles 2-4 (4-week cycle): Participants received rituximab 375 mg/m^2 IV on Day 1, mitoxantrone 10 mg/m^2 IV on Day 2, and fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 2-4. One month after completion of the above 4 cycles, participants were evaluated for tumor response (clinical and molecular evaluation). Responding participants (no progressive disease) received rituximab 375 mg/m^2 IV once weekly for a total of 4 weeks (4 total doses). Maintenance Phase: no further therapy, observation only.
Period: Induction Phase
Arm/Group | Induction Phase-Immunochemotherapy Rituximab-FND (R-FND) | Rituximab Induction, Rituximab Maintenance | Rituximab Induction, Observation Maintenance
Started | 234 | 0 | 0
Completed | 202 | 0 | 0
Not Completed | 32 | 0 | 0
Not completed — Disease progression | 14 | 0 | 0
Not completed — Adverse Event | 9 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Stable disease | 2 | 0 | 0
Not completed — Secondary neoplasia | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Follow-Up/Maintenance Phase
Arm/Group | Induction Phase-Immunochemotherapy Rituximab-FND (R-FND) | Rituximab Induction, Rituximab Maintenance | Rituximab Induction, Observation Maintenance
Started | 0 | 101 | 101
Completed | 0 | 66 | 60
Not Completed | 0 | 35 | 41
Not completed — Disease progression | 0 | 23 | 29
Not completed — Adverse Event | 0 | 3 | 1
Not completed — Death | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 4
Not completed — Relapse | 0 | 5 | 5
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) population: all participants who were randomized to the maintenance or observation arm. IP population: all enrolled participants who started the induction phase (Months 1-8 of the study)
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab Induction, Rituximab Maintenance | Rituximab Induction, Observation Maintenance | Total
Number analyzed (Participants) | 101 | 101 | 202
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [64 to 70] | 65 [62 to 69] | 66 [63 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 56 | 120
  Male | 37 | 45 | 82

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression or Death
Description: PFS from randomization was measured from the date of randomization to the date of documented disease progression, relapse, or death from any cause. PFS function was estimated using Kaplan-Meier product-limit method. Responding participants and participants who were lost to follow up were censored at their last assessment date.
Time Frame: 12, 24, and 34 months
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Induction, Rituximab Maintenance | Rituximab Induction, Observation Maintenance
Number analyzed (Participants) | 101 | 101
percentage of participants | 29.7 | 34.7
Statistical Analysis 1: Comparison: Rituximab Induction, Rituximab Maintenance vs Rituximab Induction, Observation Maintenance; Difference between treatment arms; Test type: Superiority or Other; p = 0.254, Log Rank

2. Secondary Outcome: Percentage of Participants Estimated to be Free of Progression at 12, 24, and 36 Months
Description: PFS from enrollment was measured from the date of enrollment to the date of disease progression, relapse, or death from any cause. Responding participants and participants who were lost to follow-up were censored at their last assessment date. Estimates of PFS function were made with the Kaplan-Meier product-limit method.
Time Frame: 12, 24, and 36 months
Population: IP population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Rituximab Induction: Induction Phase Cycle 1 (4-week cycle): Participants received mitoxantrone 10 mg/m^2 IV on Day 1, fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 1-3, and rituximab 375 mg/m^2 on Day 8. Induction Phase Cycles 2-4 (4-week cycle): Participants received rituximab 375 mg/m^2 IV on Day 1, mitoxantrone 10 mg/m^2 IV on Day 2, and fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 2-4. One month after completion of the above 4 cycles, participants were evaluated for tumor response (clinical and molecular evaluation). Responding participants (no progressive disease) received rituximab 375 mg/m^2 IV once weekly for a total of 4 weeks (4 total doses). Maintenance Phase: 3 months after induction treatment (Month 9), participants who showed at least a partial response after induction treatment received either no therapy (observation) or rituximab 375 mg/m^2 IV on Day 1. Doses were repeated every 2 months for a total of 4 doses.
Arm/Group | Rituximab Induction
Number analyzed (Participants) | 234
percentage of participants
  12 months | 90.1 [85.5 to 93.3]
  24 months | 77.8 [71.8 to 82.6]
  36 months | 65.7 [59.2 to 71.5]

3. Secondary Outcome: Disease-Free Survival (DFS) From Randomization - Percentage of Participants Disease Free at 12, 24, and 36 Months
Description: DFS was defined for all participants who achieved a complete response (CR) or unconfirmed CR (CRu) at Month 3 or later, after the completion of induction phase and was measured from the time of randomization to the date of relapse or death as a result of lymphoma or acute toxicity of treatment. Participants without relapse were censored at their last assessment date. Estimates of DFS were made using Kaplan-Meier product-limit method.
Time Frame: 12, 24, and 36 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab Induction, Rituximab Maintenance | Rituximab Induction, Observation Maintenance
Number analyzed (Participants) | 101 | 101
percentage of participants
  12 months | 93.0 [85.8 to 96.6] | 82.5 [73.4 to 88.8]
  24 months | 82.7 [73.7 to 88.9] | 68.9 [58.7 to 77.2]
  36 months | 69.2 [57.9 to 78.1] | 62.3 [51.2 to 71.5]
Statistical Analysis 1: Comparison: Rituximab Induction, Rituximab Maintenance vs Rituximab Induction, Observation Maintenance; Test type: Superiority or Other; p = 0.105, Cox proportional-hazards — Overall DFS; Adjusted for randomization stratum and the known prognostic factors; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.31 to 1.12]

4. Secondary Outcome: Overall Survival (OS) From Randomization - Percentage of Participants Estimated to be Alive at 12, 24, and 34 Months
Description: OS from randomization was defined as the date of randomization to the date of death from any cause. Participants still alive at the time of the final analysis were censored at the date of the last contact. Estimates of the OS function were made by the Kaplan-Meier product-limit method.
Time Frame: 12, 24, and 34 months
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Rituximab Induction, Rituximab Maintenance: Rituximab Induction, Rituximab Maintenance Induction Phase Cycle 1 (4-week cycle): Participants received mitoxantrone 10 mg/m^2 IV on Day 1, fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 1-3, and rituximab 375 mg/m^2 on Day 8. Induction Phase Cycles 2-4 (4-week cycle): Participants received rituximab 375 mg/m^2 IV on Day 1, mitoxantrone 10 mg/m^2 IV on Day 2, and fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 2-4. One month after completion of the above 4 cycles, participants were evaluated for tumor response (clinical and molecular evaluation). Responding participants (no progressive disease) received rituximab 375 mg/m^2 IV once weekly for a total of 4 weeks (4 total doses). Maintenance Phase: 3 months after induction treatment (Month 9), participants who showed at least a partial response after induction treatment received rituximab 375 mg/m^2 IV on Day 1. Doses were repeated every 2 months for a total of 4 doses.
Arm/Group | Rituximab Induction, Rituximab Maintenance | Rituximab Induction, Observation Maintenance
Number analyzed (Participants) | 101 | 101
percentage of participants
  12 months | 97.0 [91.0 to 99.0] | 100 [NA to NA] — No participants had an event, therefore 95 percent (%) confidence interval (CI) could not be determined.
  24 months | 96.0 [89.7 to 98.5] | 96.9 [90.6 to 99.0]
  34 months | 96.0 [89.7 to 98.5] | 95.8 [89.2 to 98.4]
Statistical Analysis 1: Comparison: Rituximab Induction, Rituximab Maintenance vs Rituximab Induction, Observation Maintenance; Test type: Superiority or Other; p = 0.751, Log Rank

5. Secondary Outcome: Overall Survival (OS) From Randomization - Percentage of Participants With Death
Description: as for outcome 4
Time Frame: 12, 24, and 34 months
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Induction, Rituximab Maintenance | Rituximab Induction, Observation Maintenance
Number analyzed (Participants) | 101 | 101
percentage of participants | 5.0 | 4.0
Statistical Analysis 1: Comparison: Rituximab Induction, Rituximab Maintenance vs Rituximab Induction, Observation Maintenance; Test type: Superiority or Other; p = 0.751, Log Rank

6. Secondary Outcome: OS From Enrollment - Percentage of Participants Estimated to be Alive at 12, 24, and 36 Months
Description: OS from enrollment was defined as the date of enrollment to the date of death from any cause. Participants still alive at the time of the final analysis were censored at the date of the last contact. Estimates of the OS function were made by the Kaplan-Meier product-limit method.
Time Frame: 12, 24, and 36 months
Population: IP population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab Induction, Rituximab Maintenance
Number analyzed (Participants) | 234
percentage of participants
  12 months | 94.9 [91.1 to 97.0]
  24 months | 92.7 [88.4 to 95.4]
  36 months | 89.5 [84.8 to 92.9]

7. Primary Outcome: PFS Randomization- Percentage of Participants Estimated to be Free of Progression at 12, 24, and 34 Months
Description: PFS from randomization was measured from the date of randomization to the date of documented disease progression, relapse, or death from any cause. Responding participants and participants who were lost to follow-up were censored at their last assessment date. PFS was estimated using Kaplan-Meier methods.
Time Frame: 12, 24, and 34 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab Induction, Rituximab Maintenance | Rituximab Induction, Observation Maintenance
Number analyzed (Participants) | 101 | 101
percentage of participants
  12 months | 92.0 [84.7 to 95.9] | 82.5 [73.4 to 88.8]
  24 months | 81.0 [71.8 to 87.4] | 68.9 [58.7 to 77.2]
  34 months | 70.4 [60.2 to 78.4] | 62.3 [51.2 to 71.5]
Statistical Analysis 1: Comparison: Rituximab Induction, Rituximab Maintenance vs Rituximab Induction, Observation Maintenance; Analysis of overall PFS with Cox proportional-hazards model adjusted for the randomization stratum and the known prognostic factors; Test type: Superiority or Other; p = 0.079, Cox proportional-hazards; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.38 to 1.05]

8. Secondary Outcome: Percentage of Participants With a Response During the Induction Phase
Description: Participants without a response assessment (due to any reasons) were considered as non-responders.
Time Frame: Months 1 to 8
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Induction, Rituximab Maintenance | Rituximab Induction, Observation Maintenance
Number analyzed (Participants) | 101 | 101
percentage of participants
  Complete remission (CR/CRu) | 79.2 | 79.2
  Partial remission | 19.8 | 19.8
  Stable disease | 1.0 | 0.0
  Progression disease | 0.0 | 0.0
  Missing | 0.0 | 1.0

9. Secondary Outcome: Percentage of Participants With a Molecular Response in the Induction Phase
Description: Molecular responders were defined as the proportion of CR/CRu participants with a positive bcl-2/IgH (non-Hodgkin's Lymphoma [NHL] marker) at baseline, whose laboratory values were undetectable after treatment.
Time Frame: Months 5 and 8
Population: IP population; only participants with a positive bcl-2/IgH (NHL marker) at baseline were included in the analysis.
Measure: Number; unit: percentage of participants
Groups:
- Rituximab Induction, Rituximab Maintenance: Induction Phase Cycle 1 (4-week cycle): Participants received mitoxantrone 10 mg/m^2 IV on Day 1, fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 1-3, and rituximab 375 mg/m^2 on Day 8. Induction Phase Cycles 2-4 (4-week cycle): Participants received rituximab 375 mg/m^2 IV on Day 1, mitoxantrone 10 mg/m^2 IV on Day 2, and fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 2-4. One month after completion of the above 4 cycles, participants were evaluated for tumor response (clinical and molecular evaluation). Responding participants (no progressive disease) received rituximab 375 mg/m^2 IV once weekly for a total of 4 weeks (4 total doses). Maintenance Phase: 3 months after induction treatment (Month 9), participants who showed at least a partial response after induction treatment received either no treatment (observation) or rituximab 375 mg/m^2 IV on Day 1. Doses were repeated every 2 months for a total of 4 doses.
Arm/Group | Rituximab Induction, Rituximab Maintenance
Number analyzed (Participants) | 118
percentage of participants
  Month 5 | 36.4
  Month 8 | 58.5

10. Secondary Outcome: Duration of Response Using a Traditional Approach - Percentage of Participants Estimated to Have a Sustained Response at 12, 24, and 34 Months
Description: Duration of response (DOR) was defined for all participants who achieved a response (CR, CRu, and PR) at Month 3 or later, after the completion of induction phase and was measured from the date of randomization until the date of progression, relapse, or death as a result of follicular lymphoma (FL). Participants without relapse, progression, or death for causes other than FL were censored at their last assessment date. Analyses on this endpoint were performed with two different approaches. For the traditional approach, duration of response was estimated as the proportion of participants alive without progression or relapse of disease with the Kaplan-Meier method.
Time Frame: Months 12, 24, and 34
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab Induction, Rituximab Maintenance | Rituximab Induction, Observation Maintenance
Number analyzed (Participants) | 100 | 99
percentage of participants
  12 Months | 93.9 [86.9 to 97.2] | 82.3 [73.1 to 88.6]
  24 Months | 83.6 [74.6 to 89.6] | 68.6 [58.3 to 76.9]
  34 Months | 69.9 [58.5 to 78.7] | 61.9 [50.9 to 71.2]
Statistical Analysis 1: Comparison: Rituximab Induction, Rituximab Maintenance vs Rituximab Induction, Observation Maintenance; Test type: Superiority or Other; p = 0.103, Regression, Cox — Univariate analysis; Cox model stratified for the stratification groups; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.40 to 1.09]
Statistical Analysis 2: Comparison: Rituximab Induction, Rituximab Maintenance vs Rituximab Induction, Observation Maintenance; Test type: Superiority or Other; p = 0.071, Regression, Cox — Multivariate analysis; Adjusted for stratification group, age, sex, Eastern Cooperative Oncology Group Performance Status, FL International prognostic index (FLIPI) score; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.37 to 1.04]

11. Secondary Outcome: Duration of Response Using the Competing Risk Approach - Cumulative Percentage of Participants With Progression, Relapse or Death as a Result of FL at 12, 24, and 34 Months
Description: DOR was defined for all participants who achieved a response (CR, CRu, and PR) at Month 3 or later, after the completion of induction phase and was measured from the date of randomization until the date of progression, relapse, or death as a result of FL. Participants without relapse, progression, or death for causes other than FL were censored at their last assessment date. Analyses on this endpoint were performed with two different approaches. For the competing risk approach, deaths for causes other than FL were considered as competing events. DOR was estimated with the cumulative incidence of progression, relapse, or death as a result of FL.
Time Frame: Months 12, 24, and 34
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab Induction, Rituximab Maintenance | Rituximab Induction, Observation Maintenance
Number analyzed (Participants) | 100 | 99
percentage of participants
  12 Months | 6.1 [1.3 to 10.8] | 17.7 [10.0 to 25.3]
  24 Months | 16.2 [8.9 to 23.5] | 31.4 [22.0 to 40.8]
  34 Months | 29.5 [19.5 to 39.6] | 38.0 [27.8 to 48.3]
Statistical Analysis 1: Comparison: Rituximab Induction, Rituximab Maintenance vs Rituximab Induction, Observation Maintenance; Test type: Superiority or Other; p = 0.084, Fine and Gray model — Univariate analysis; Fine and Gray model stratified for the stratification groups; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.39 to 1.06]
Statistical Analysis 2: Comparison: Rituximab Induction, Rituximab Maintenance vs Rituximab Induction, Observation Maintenance; Test type: Superiority or Other; p = 0.052, Fine and Gray model; Fine and Gray model adjusted for stratification group, age, sex, Eastern Cooperative Oncology Group Performance Status, and FLIPI score; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.38 to 1.00]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported up to Month 15.
Description: Analyses were performed including all patients receiving at least one dose of planned therapy, both on IP and ITT population. One participant in the Induction Phase did not receive any study drug was not included in the analysis.
Groups:
- Rituximab Induction (Induction Phase Only): Rituximab Induction, Rituximab Maintenance Induction Phase Cycle 1 (4-week cycle): Participants received mitoxantrone 10 mg/m^2 IV on Day 1, fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 1-3, and rituximab 375 mg/m^2 on Day 8. Induction Phase Cycles 2-4 (4-week cycle): Participants received rituximab 375 mg/m^2 IV on Day 1, mitoxantrone 10 mg/m^2 IV on Day 2, and fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 2-4. One month after completion of the above 4 cycles, participants were evaluated for tumor response (clinical and molecular evaluation). Responding participants (no progressive disease) received rituximab 375 mg/m^2 IV once weekly for a total of 4 weeks (4 total doses).
- Rituximab Induction, Rituximab Maintenance (Follow-up Phase): Rituximab Induction, Rituximab Maintenance Induction Phase Cycle 1 (4-week cycle): Participants received mitoxantrone 10 mg/m^2 IV on Day 1, fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 1-3, and rituximab 375 mg/m^2 on Day 8. Induction Phase Cycles 2-4 (4-week cycle): Participants received rituximab 375 mg/m^2 IV on Day 1, mitoxantrone 10 mg/m^2 IV on Day 2, and fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 2-4. One month after completion of the above 4 cycles, participants were evaluated for tumor response (clinical and molecular evaluation). Responding participants (no progressive disease) received rituximab 375 mg/m^2 IV once weekly for a total of 4 weeks (4 total doses). Maintenance Phase: 3 months after induction treatment (Month 9), participants who showed at least a partial response after induction treatment received rituximab 375 mg/m^2 IV on Day 1. Doses were repeated every 2 months for a total of 4 doses.
- Rituximab Induction, Observation Maintenance (Follow-up Phase): Induction Phase Cycle 1 (4-week cycle): Participants received mitoxantrone 10 mg/m^2 IV on Day 1, fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 1-3, and rituximab 375 mg/m^2 on Day 8. Induction Phase Cycles 2-4 (4-week cycle): Participants received rituximab 375 mg/m^2 IV on Day 1, mitoxantrone 10 mg/m^2 IV on Day 2, and fludarabine 25 mg/m^2 IV and dexamethasone 10 mg IV on Days 2-4. One month after completion of the above 4 cycles, participants were evaluated for tumor response (clinical and molecular evaluation). Responding participants (no progressive disease) received rituximab 375 mg/m^2 IV once weekly for a total of 4 weeks (4 total doses). Maintenance Phase: no further therapy, observation only.
Arm/Group | Rituximab Induction (Induction Phase Only) | Rituximab Induction, Rituximab Maintenance (Follow-up Phase) | Rituximab Induction, Observation Maintenance (Follow-up Phase)
Serious Adverse Events (participants affected / at risk) | 19/233 | 19/101 | 17/101
Other Adverse Events (participants affected / at risk) | 230/233 | 73/101 | 55/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Induction (Induction Phase Only) (N=233) | Rituximab Induction, Rituximab Maintenance (Follow-up Phase) (N=101) | Rituximab Induction, Observation Maintenance (Follow-up Phase) (N=101)
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Pyrexia (Immune system disorders) | 2 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0
Febrile neutropenia (Infections and infestations) | 2 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 1 | 2
Pneumonitis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Spinal compression fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Pulmonary embolism (Vascular disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac ablation (Cardiac disorders) | 0 | 1 | 0
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Diabetic vascular disorder (Endocrine disorders) | 0 | 1 | 0
Cholecystitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 2
Septic shock (Infections and infestations) | 0 | 1 | 0
Transient ischaemic shock (Nervous system disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 2
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1
Cholelithiasis (Gastrointestinal disorders) | 0 | 0 | 3
Femur fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hip arthroplasty (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Upper limb fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Cataract operation (Eye disorders) | 0 | 0 | 1
Ovarian adenoma (Reproductive system and breast disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Induction (Induction Phase Only) (N=233) | Rituximab Induction, Rituximab Maintenance (Follow-up Phase) (N=101) | Rituximab Induction, Observation Maintenance (Follow-up Phase) (N=101)
Bronchospasm (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 2 | 0 | 0
Escherichia infection (Infections and infestations) | 1 | 1 | 0
Fungal infection (Infections and infestations) | 2 | 0 | 0
Genitourinary tract infection (Infections and infestations) | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 6 | 0 | 0
Herpes zoster (Infections and infestations) | 4 | 2 | 3
Klebsiella infection (Infections and infestations) | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 0
Prostate infection (Infections and infestations) | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 2 | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Vaginal candidiasis (Infections and infestations) | 1 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral DNA test positive (Infections and infestations) | 1 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Pneumonitis (Infections and infestations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 3 | 1 | 7
Lung infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngeal disorder (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 2 | 2
Rhinitis (Infections and infestations) | 0 | 4 | 2
Influenza (Infections and infestations) | 7 | 5 | 9
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Choking sensation (Gastrointestinal disorders) | 2 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 6 | 0 | 1
Hypersensitivity (Immune system disorders) | 11 | 0 | 1
Edema (General disorders) | 11 | 0 | 0
Hyperpyrexia (General disorders) | 1 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 1
Infusion related reaction (General disorders) | 2 | 0 | 0
Oedema (General disorders) | 2 | 0 | 2
Oedema peripheral (General disorders) | 7 | 2 | 0
Pharyngeal oedema (General disorders) | 2 | 8 | 0
Pyrexia (General disorders) | 44 | 8 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Skin (Skin and subcutaneous tissue disorders) | 8 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Neck mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin infection (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Altered hearing (Ear and labyrinth disorders) | 2 | 0 | 0
Deafness (Ear and labyrinth disorders) | 2 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 103 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 225 | 16 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 120 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 5 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 2 | 0
Ischaemia (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 7 | 2 | 1
Hypotension (Vascular disorders) | 3 | 1 | 1
Pulse pressure increased (Vascular disorders) | 1 | 0 | 0
Asthenia (General disorders) | 16 | 4 | 5
Asthenia/fatigue (General disorders) | 57 | 0 | 0
Chills (General disorders) | 4 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 1
Oedema mucosal (General disorders) | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 6 | 1 | 0
Feeling hot (General disorders) | 1 | 0 | 0
Diabetes mellitus (Endocrine disorders) | 2 | 0 | 1
Diabetic vascular disorder (Endocrine disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 16 | 0 | 0
Insomnia (Psychiatric disorders) | 7 | 1 | 0
Weight increased (Investigations) | 2 | 0 | 0
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Thyroiditis chronic (Endocrine disorders) | 1 | 0 | 0
Abdominal ridigity (Gastrointestinal disorders) | 1 | 0 | 0
Anal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 24 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 23 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 5 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 2 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 43 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1 | 0
Pulpitis dental (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 23 | 2 | 0
Vomiting (Gastrointestinal disorders) | 8 | 2 | 0
Furuncle (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Anal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0
Helicobacter pylori identification test positive (Infections and infestations) | 0 | 1 | 0
Hepatitis viral (Infections and infestations) | 0 | 1 | 0
Pancreatic disorder (Gastrointestinal disorders) | 0 | 1 | 0
Polyp colorectal (Gastrointestinal disorders) | 0 | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 10 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 12 | 2 | 1
Blood amylase increased (Investigations) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1
Beta 2 microglobulin increased (Investigations) | 0 | 1 | 1
Blood immunoglobulin A decreased (Investigations) | 0 | 0 | 1
Blood immunoglobulin G decreased (Investigations) | 0 | 0 | 1
Blood immunoglobulin M decreased (Investigations) | 1 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 4 | 2 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase (Investigations) | 1 | 1 | 0
Hyperkalaemia (Investigations) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 1 | 0 | 0
Transaminases abnormal (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase (Investigations) | 0 | 1 | 0
Blood amylase (Investigations) | 0 | 1 | 0
Alanine aminotransferase (Investigations) | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0
Haemoglobin increaed (Investigations) | 0 | 1 | 0
Fistula (General disorders) | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Ejection fracture decreased (Cardiac disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Aptyalism (Endocrine disorders) | 0 | 0 | 1
Total bile acids increased (Investigations) | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 0 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 0 | 0
Chest pain (General disorders) | 4 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1
Pelvic pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pain (General disorders) | 31 | 0 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bone density increased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Movement disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 1 | 3
Dysuria (Renal and urinary disorders) | 4 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 13 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 0
Facial palsy (Nervous system disorders) | 1 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0
Neuropathy (Nervous system disorders) | 1 | 1 | 0
Neuropathy: motor (Nervous system disorders) | 5 | 0 | 0
Neuropathy: sensory (Nervous system disorders) | 9 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0
Paraesthesia oral (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 7 | 3 | 0
Migraine (Nervous system disorders) | 2 | 0 | 0
Amnesia (Psychiatric disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vagotomy (Nervous system disorders) | 1 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 0 | 0
Phlebitis (Vascular disorders) | 2 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Blood pressure increased (Vascular disorders) | 0 | 0 | 1
Carotid artery stenosis (Vascular disorders) | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign prostatic hyperplasia (Renal and urinary disorders) | 1 | 0 | 1
Cystitis (Infections and infestations) | 5 | 1 | 4
Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1
Urinary tract disorder (Renal and urinary disorders) | 1 | 0 | 1
Prostate examination abnormal (Renal and urinary disorders) | 0 | 0 | 1
Vaginal burning sensation (Reproductive system and breast disorders) | 0 | 1 | 0
Bronchitis chronic (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.